CLINICAL TRIAL: NCT02344095
Title: A Randomized Phase 1 Trial Evaluating the Safety of Weekly Paclitaxel With Oncothermia and Weekly cisPlatin With Oncothermia in Patients With Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: A Trial of Weekly Paclitaxel With Oncothermia and Weekly cisPlatin With Oncothermia in Patients With Recurrent or Persistent Ovarian Cancer
Acronym: POPOPO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yong Beom Kim, MD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGOG3030
Record Dates: First submitted 2014-11-01; First posted 2015-01-22 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Epithelial Ovarian Carcinoma; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
Keywords: recurrent, persistent
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- weekly paclitaxel with oncothermia (Experimental): Paclitaxel group are treated with weekly paclitaxel and oncothermia for 4-cycles.
  Interventions: Drug: weekly paclitaxel; Device: oncothermia
- weekly cisplatin with oncothermia (Experimental): Cisplatin group are treated with weekly cisplatin and oncothermia for 4-cycles.
  Interventions: Drug: weekly cisplatin; Device: oncothermia

INTERVENTIONS:
Drug: weekly paclitaxel — Patients are treated with weekly paclitaxel 70mg/m2 (IV) on day 1, 8, and 15 at an intervals of 4 weeks
  Arms: weekly paclitaxel with oncothermia
Drug: weekly cisplatin — Patients are treated with weekly cisplatin 40mg/m2 (IV) on day 1, 8, and 15 at an intervals of 4 weeks.
  Arms: weekly cisplatin with oncothermia
Device: oncothermia — Thermotherapy is performed by applying oncothermia (EHY 2000) probe on the part of body where tumor is located and delivering energy. It is performed on day 1, 4, 8, 11, 15, 18, 21, and 24 (8 times in total every cycle). Oncothermia can be performed a day earlier than scheduled day or a day later than scheduled day. With tumors at multiple sites, oncothermia is performed several times changing sites that apply probe and type of probes.
  - It takes 60 minutes to treat a site for oncothermia. Energy is gradually increased from 60W to 140W.

SUMMARY:
The investigators aimed to evaluate the safety of weekly paclitaxel with oncothermia and weekly cisplatin with oncothermia in patients with recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma. This trial is a randomized phase 1 trial. The investigators planned to perform it for 1 year. In this trial, a total of 12 patients with recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma are randomly assigned to either a paclitaxel or cisplatin group in ratio of 1 to 1. Paclitaxel group are treated with weekly paclitaxel and oncothermia. Cisplatin group are treated with weekly cisplatin and oncothermia. In each group, limiting toxicity is evaluated after treating 3 patients for 4-cycles. Primary endpoint is occurrence of limiting toxicity. Secondary endpoints are response rate, progression-free survival, overall-survival, quality of life, pain, fatigue and compliance rate.

DETAILED DESCRIPTION:
This trial is a randomized phase 1 trial. We planned to perform it for 1 year. Subjects of study are patients diagnosed as recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma. The number of subjects of study is 12 patients (If patients cannot be assessed, they can be replaced with new patients). All subjects who were randomly assigned, are treated with weekly paclitaxel or weekly cisplatin. In paclitaxel group, patients are treated with weekly paclitaxel 70mg/m2 (IV) on day 1, 8, and 15 at an intervals of 4 weeks. In cisplatin group, patients are treated with weekly cisplatin 40mg/m2 (IV) on day 1, 8, and 15 at an intervals of 4 weeks. Thermotherapy is performed by applying oncothermia (EHY 2000) probe on the part of body where tumor is located and delivering energy. It is performed on day 1, 4, 8, 11, 15, 18, 21, and 24 (8 times in total every cycle). Oncothermia can be performed a day earlier than scheduled day or a day later than scheduled day. It takes 60 minutes to treat a site for oncothermia. Energy is gradually increased from 60W to 140W. With tumors at multiple sites, oncothermia is performed several times changing sites that apply probe and type of probes. Oncothermia is performed for 60 minutes per each application. Patients with recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma are randomly assigned to either a paclitaxel or cisplatin group in ratio of 1 to 1. Paclitaxel group are treated with weekly paclitaxel and oncothermia. Cisplatin group are treated with weekly cisplatin and oncothermia. In each group, limiting toxicity is evaluated after treating 3 patients for 4-cycles. In group that limiting toxicity occur in the rate equal to or less than 1 patient, limiting toxicity is evaluated after treating 3 additional patients for 4-cycles. When limiting toxicity occur in the rate equal to or less than one of six assessable patients, it is considered that the specific therapy is safe enough to be used in phase 2 trial. Primary endpoint is occurrence of limiting toxicity. Secondary endpoints are response rate, progression-free survival, overall-survival, quality of life, toxicity, pain, fatigue and compliance rate. Patients visit twice a week until 4-cycles are completed or progression of disease is confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma (At the first diagnosis, pathologic findings should be confirmed.)
* Response assessments that are possible by using radiologic tests or tumor markers
* The number of chemotherapeutic regimens that were previously used ≤ 2
* Adequate hematologic, hepatic, and renal functions
* ECOG performance status 0 - 2

Exclusion Criteria:

* Recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma that are located on the part of body where it is impossible to deliver energy by using oncothermia (EHY 2000) probe
* Neurotoxicity ≥ grade 2
* Pacemaker user
* Large metal materials such as artificial joint that are kept in the body
* Recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma that are located on the part of body where got previously radiation therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of limiting toxicity | 8 cycles up to 1 year
  When limiting toxicity occur in the rate equal to or more than two of six assessable patients, study would be closed.

SECONDARY OUTCOMES:
response rate | 8 cycles up to 1 year
  When limiting toxicity occur in the rate equal to or more than two of six assessable patients, study would be closed.
progression-free survival | 8 cycles up to 1 year
  When limiting toxicity occur in the rate equal to or more than two of six assessable patients, study would be closed.
overall-survival | 8 cycles up to 1 year
  When limiting toxicity occur in the rate equal to or more than two of six assessable patients, study would be closed.
quality of life, assessed with the Korean version of WHO Quality of Life-BREF (WHOQOL-BREF). | 8 cycles up to 1 year
  When limiting toxicity occur in the rate equal to or more than two of six assessable patients, study would be closed. Quality of life would be assessed with the Korean version of WHO Quality of Life-BREF (WHOQOL-BREF).
pain, assessed with the Korean version of the brief pain inventory (BPI). | 8 cycles up to 1 year
  When limiting toxicity occur in the rate equal to or more than two of six assessable patients, study would be closed. Pain would be assessed with the Korean version of the brief pain inventory (BPI).
fatigue, assessed with the Korean version of the Brief Fatigue Inventory (BFI). | 8 cycles up to 1 year
  When limiting toxicity occur in the rate equal to or more than two of six assessable patients, study would be closed. Fatigue would be assessed with the Korean version of the Brief Fatigue Inventory (BFI).
compliance rate | 8 cycles up to 1 year
  When limiting toxicity occur in the rate equal to or more than two of six assessable patients, study would be closed. Compliance rate would be assessed with the number of patients that are dropped out from current clinical trial based on other reasons instead of disease. It would be recorded as compliance rate = the number of patients that are dropped out due to other reasons/the number of total patients · 100 (%)

CONTACTS AND LOCATIONS:
Overall Officials: Kidong kim, MD, Study Director — Seoul National University Bundang Hospital,Gyeongg-ido,Repub
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim K, Kim JH, Kim SC, Kim YB, Nam BH, No JH, Cho H, Ju W, Suh DH, Kim YH. Modulated electro-hyperthermia with weekly paclitaxel or cisplatin in patients with recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma: The KGOG 3030 trial. Exp Ther Med. 2021 Jul;22(1):787. doi: 10.3892/etm.2021.10219. Epub 2021 May 21. PMID 34055086